CLINICAL TRIAL: NCT04427410
Title: The Relationship Between Oxytocin Level Measured During Pregnancy and Postpartum Depression Symptoms
Brief Title: The Relationship Between Oxytocin Level and Postpartum Depression
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Collaborators: Ayseren Cevik (Unknown)
Responsible Party: Principal Investigator, Sultan Alan, Associate Professor Dr, Cukurova University
Other Study IDs: TYL-2019-12476
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Oxytocin Deficiency; Postpartum Depression; Prenatal Stress
Keywords: oxytocin; Postpartum Depression; oxytocin and depression
MeSH Terms: conditions — Depression, Postpartum; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pregnancy
  Interventions: Diagnostic Test: Salivary test
- postpartum
  Interventions: Diagnostic Test: Salivary test

INTERVENTIONS:
Diagnostic Test: Salivary test — Salivary test for measured of oxytocin levels
  Other Names: survey application

SUMMARY:
There are studies in the literature that associate oxytocin level with postpartum depression. This study was carried out to investigate the relationship between oxytocin levels measured during pregnancy and postpartum depression symptoms.

DETAILED DESCRIPTION:
Introduction and purpose: There are studies in the literature that associate oxytocin level with postpartum depression. This study was carried out to investigate the relationship between oxytocin levels measured during pregnancy and postpartum depression symptoms.

Method: The study was conducted with 70 women who met the research criteria. Data collection was done in two interviews. The first meeting is 30-38 at the week of gestation, the second interview is 4-12 at the week of postpartum. It was done between weeks. In each interview, a data collection form was applied first and then a saliva sample was taken. Data collection form; The questions prepared by the researchers consisted of the Edinburgh Postnatal Depression Scale (EPDS) and Beck Depression Inventory (BDI). The data were analyzed using SPSS 22.0 program and the significance value was taken as p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, and having a pregnancy of 30 weeks or more

Exclusion Criteria:

* previous mental illness history, miscarriage or stillbirth history, multiple pregnancy, fetal malformation, antidepressant or anxiolytic drug use, existing chronic disease,preterm labor is the development of maternal or neonatal complications at birth, hospitalization in the neonatal intensive care unit or congenital disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnancy and postpartum period
Study Population: Based on the study conducted by Eapen et al. (2014), for the relationship between oxytocin and postpartum depression symptoms, based on the correlation coefficient for the periods during and after pregnancy; For r = -0.35, a minimum sample size of 61 with 5% error and 80% power has been determined. Since there may be a quit situation during the study, the sample size was determined as 67 by expanding it with a share of 10%.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Oxytocin levels | 3-6 month
  Oxytocin levels in pregnancy and postpartum period

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Saricam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No